CLINICAL TRIAL: NCT03842839
Title: Effect of Tiotropium on Airway Remodeling in Patients With Early Stage COPD Accessed by Optical Coherence Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Professor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCOPD-20181001
Record Dates: First submitted 2019-01-21; First posted 2019-02-15 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Airway Remodeling
MeSH Terms: conditions — Airway Remodeling | interventions — Tiotropium Bromide; Albuterol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tiotropium (0-12 month) + SABA as needed (Experimental): * During the 2 years treatment phase patients will be administered with tiotropium bromide (Spiriva) capsule 18μg once daily from baseline to the 12th months.
  * Any long acting bronchodilator will not be used from the 12 to 24 months.
  * Salbutamol sulphate aerosol (Ventolin) will be administered as concomitant medication treatment when exacerbation occurs.
  Interventions: Drug: Tiotropium Inhalation Powder [Spiriva] 0.018mg; Drug: Salbutamol sulphate aerosol (Ventolin) 0.01mg
- Tiotropium (0-24 month) + SABA as needed (Experimental): * During the 2 years treatment phase patients will be administered with tiotropium bromide (Spiriva) capsule 18μg once daily from baseline to the 24th months.
  * Salbutamol sulphate aerosol (Ventolin) will be administered as concomitant medication treatment when exacerbation occurs.
  Interventions: Drug: Tiotropium Inhalation Powder [Spiriva] 0.018mg; Drug: Salbutamol sulphate aerosol (Ventolin) 0.01mg
- SABA as needed only (Other): * During the 2 years treatment phase patients will be administered with salbutamol sulphate aerosol (Ventolin) when exacerbation occurs.
  * Any long acting bronchodilator will not be used during the 2 years treatment phase.
  Interventions: Drug: Salbutamol sulphate aerosol (Ventolin) 0.01mg

INTERVENTIONS:
Drug: Tiotropium Inhalation Powder [Spiriva] 0.018mg — Tiotropium bromide (Spiriva) capsule 18μg once daily inhaled.
  Other Names: Spiriva
  Arms: Tiotropium (0-12 month) + SABA as needed; Tiotropium (0-24 month) + SABA as needed
Drug: Salbutamol sulphate aerosol (Ventolin) 0.01mg — As needed use of salbutamol sulphate aerosol (Ventolin) when exacerbation happens
  Other Names: Ventolin

SUMMARY:
The study aims to explore the effect of tiotropium on airway remodeling by using Endobronchial Optical Coherence Tomography (EB-OCT). We enrolled patients with GOLD I stage COPD. All the patients will be divided into four groups randomly to receive SABA as needed with or without regular use of tiotropium. Changes of airway morphology (accessed by EB-OCT), pulmonary function, QOL, and SABA usage will be obtained.

ELIGIBILITY:
Key inclusion criteria

* Over 40 yrs; Male or female Diagnosed with COPD
* Pre-bronchodilator FEV1 ≥80% pred ;
* Patients must be able to perform all study related procedures

Exclusion Criteria:

* Patients with other lung diseases (such as bronchiectasis, pneumothorax, pleural effusion, airway deformation, lung surgery, etc.).
* Patients have poor compliance and are unwilling to receive medication regularly.
* Other complications of bronchoscopy or intolerance of bronchoscopy procedure.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the inner luminal area (Ai) of the 3th to 9th generation bronchi at month 24 | Ai accessed by endobronchial optical coherence tomography will be obtained at baseline, month 24.
  To evaluate the effects of Tiotropium in ameliorating airway remodeling in early stage COPD
Change from baseline in the inner luminal area (Ai) of the 3th to 9th generation bronchi at month 12 | Ai accessed by endobronchial optical coherence tomography will be obtained at month 12.
  To evaluate the effects of Tiotropium in ameliorating airway remodeling in early stage COPD

SECONDARY OUTCOMES:
Change from baseline in the airway wall area percentage (Aw%) of the 3th to 9th generation bronchi at month 12 | Aw% accessed by endobronchial optical coherence tomography will be obtained at baseline, month 12.
  To evaluate the effects of Tiotropium in ameliorating airway remodeling in early stage COPD
Change from baseline in the airway wall area percentage (Aw%) of the 3th to 9th generation bronchi at month 24 | Aw% accessed by endobronchial optical coherence tomography will be obtained at month24.
  To evaluate the effects of Tiotropium in ameliorating airway remodeling in early stage COPD
Change from baseline in trough FEV1 | Pulmonary function test will be performed at baseline, month 6, 12, 18 and 24.
  To evaluate the effects of Tiotropium in improving lung function
Change from baseline in resonant frequency (Fres) at month 6, 12, 18 and 24. | IOS will be performed at baseline, month 6, 12, 18 and 24.
  To evaluate the effects of Tiotropium in improving lung function
Change from baseline in peripheral airway resistance (R5-R20) | IOS will be performed at baseline, month 6, 12, 18 and 24.
  To evaluate the effects of Tiotropium in improving lung function
Total times of SABA usage | During the two years treatment period, times of SABA administration will be recored.
  To evaluate the times of SABA administration
Total dosage of SABA usage | During the two years treatment period, the dosage of SABA administration will be recored.
  To evaluate the dosage of SABA administration

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China